CLINICAL TRIAL: NCT02222363
Title: A Phase I Study of the Safety and Tolerability of VLX600, an Iron Chelator, in Patients With Refractory Advanced Solid Tumors
Brief Title: Study of Safety and Tolerability of VLX600, an Iron Chelator, in Patients With Refractory Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment and lack of efficacy despite the completion of several dose steps.
Sponsor: Vivolux AB (Industry)
Collaborators: Theradex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V13-11045; IND 118039 (Other: CDER/DOP2/OHOP)
Record Dates: First submitted 2014-08-15; First posted 2014-08-21 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Refractory Cancer
Keywords: Phase I; Iron chelator; Refractory advanced solid tumors; Dose escalation study; Safety and tolerability; Tumor response by RECIST 1.1; Progression-free survival; Overall survival Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — VLX600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VLX600 (Experimental): Dose of VLX600 in patients with refractory advanced solid tumors
  Interventions: Drug: VLX600

INTERVENTIONS:
Drug: VLX600 — Patients will receive a dose of VLX600 by 4-hr intravenous infusion using a central venous catheter on Days 1, 8, and 15 of each 28-day treatment cycle. There are the following dose cohorts: 10, 20, 40, 80, 160, and 210 mg VLX600. It is anticipated that patients will receive 6 treatment cycles. In the absence of unacceptable toxicity and disease progression, patients have the option of continuing treatment beyond 6 cycles, if the investigator determines that the patient may benefit further from it.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the investigational drug VLX600 in patients with refractory advanced solid tumors.

DETAILED DESCRIPTION:
This Phase I, open label dose escalation study of VLX600 in patients with refractory advanced solid tumors will determine the safety profile and maximum tolerated dose (MTD) of VLX600 when administered by intravenous infusion on Days 1, 8, and 15 of each 28-day treatment cycle. Dose escalation will proceed according to the standard "3 + 3" design using doubling doses. The doses are: 10, 20, 40, 80, 160, and 210 mg VLX600.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women greater than or equal to 18 years of age.
2. Histologic evidence of advanced solid tumors (excluding central nervous system (CNS) primary tumors) non-resectable, refractory to standard therapies, or patient cannot receive or refuses standard therapy.
3. Solid tumors measurable according to RECIST 1.1 or solid tumors not measurable according to RECIST 1.1, but which express tumor markers (e.g., prostate cancer with prostate specific antigen (PSA) expression or ovarian cancer with cancer antigen-125 (CA-125) expression) are eligible.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
5. Must have the following laboratory values, obtained less than or equal to 7 days prior to registration:

   * Absolute neutrophil count (ANC) greater than or equal to 1500/µL
   * Platelet (PLT) count greater than or equal to 100,000/µL
   * Total bilirubin less than 1.5 x upper normal limit (UNL)
   * Aspartate aminotransferase (AST) (SGOT) less than or equal to 3 x UNL
   * Creatinine less than 1.5 x UNL
6. Women of childbearing potential must have a negative serum pregnancy test less than or equal to 7 days prior to registration.
7. Life expectancy greater than 12 weeks.
8. Must provide written informed consent.
9. Must be willing to return to Mayo Clinic enrolling institution for follow-up.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, diabetes mellitus, seizure disorder or psychiatric illness/social situations that would limit compliance with study requirements.
2. Treatment with any of the following prior therapies:

   * Chemotherapy less than or equal to 4 weeks prior to registration
   * Mitomycin C/nitrosoureas less than or equal to 6 weeks prior to registration
   * Immunotherapy less than or equal to 4 weeks prior to registration
   * Biologic therapy less than or equal to 4 weeks prior to registration
   * Radiation therapy less than or equal to 4 weeks prior to registration
   * Non-cytotoxic therapy less than or equal to 5 half-lives prior to registration
3. Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment.
4. Major surgery less than 28 days prior to study entry.
5. Active other malignancy, except non-melanoma skin cancer or carcinoma-in-situ (e.g., of cervix, breast, prostate). If there is a history of prior malignancy, patient must not be receiving other specific treatment (other than hormonal therapy) for the cancer.
6. CNS metastases if not previously treated and stable for at least 2 months per imaging and clinical assessment.
7. Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

   * Pregnant women
   * Nursing women
   * Men or women of childbearing potential unwilling to employ adequate contraception
8. Other concurrent chemotherapy, immunotherapy, radiotherapy, any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation) or receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
9. Cardiac issues consisting of either symptomatic congestive heart failure (NYHA Class II or higher), unstable angina pectoris, myocardial infarction within 6 months, and/or cardiac arrhythmia, including atrial fibrillation (which is symptomatic or requires treatment).
10. Corrected QT interval (QTc) interval greater than 450 msec (males) or greater than 470 msec (females).
11. Immunocompromised patients (other than that related to the use of corticosteroids) including patients with a known history of human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
12. Clinically relevant retinal abnormalities as per the medical history or ophthalmologic findings in the pretreatment evaluation (e.g., retinitis pigmentosa or macular degeneration).
13. History of thromboembolism within the past 5 years, history of catheter-related thrombophlebitis or other clinically significant thrombophlebitis are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse event (AE) profile | AEs are assessed from first treatment day through at least 30 days after last treatment.
Determination of the maximum tolerated dose (MTD) of VLX600 | MTD will be determined during dose escalation phase of study, up to one year.
Determination of the recommended Phase II dose (RPTD) of VLX600 | Determination of RPTD will be based on adverse event profile, up to one year.

SECONDARY OUTCOMES:
Description of the tumor response to VLX600 treatment | Tumor response will be evaluated by CT scans or MRI at pre-treatment baseline and on Cycle 2 Day 28, then after every 8 weeks, and then at off-study (if greater than 4 weeks since prior tumor assessment).
  Tumor response will be determined using CT scans or magnetic resonance imaging (MRI) at pre-treatment, Cycle 2 Day 28, at every 8 weeks thereafter, and at off-study (if a scan has not been performed within the last prior 4 weeks). Patients in the MTD confirmation cohort only will have a pre-treatment baseline positron emission tomography- computerized tomography (PET-CT) scan and then at Cycle 2 Day 28. Tumor response will be determined by Response Criteria in Solid Tumors (RECIST) version 1.1. In patients with disease not measurable by RECIST 1.1, blood samples for biomarkers of tumor response will be collected at pre-treatment baseline and then after every 8 weeks.
Description of progression-free survival | Progression-free survival is calculated from date of first treatment until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 200 days (through 6 treatment cycles).
Description of the pharmacokinetics (PK) of VLX600 | PK assessed in Cycle 1 only. Day 1: pre-dose, 15, 30, 60 min, and 2, 4, 4.25, 4.5, 5, 8 hrs post start of infusion. Day 2: 24 hr post-start of infusion. Day 8: pre-dose, Day 15 (same as Day 1), Day 16: 24 hr post-start of infusion, and Day 22: pre-dose
  Blood samples will be collected for PK analysis at the specified time points in Cycle 1 only.
Description of overall survival. | Overall survival will be determined from date of first study treatment until death due to any cause, up to 72 weeks (duration of study).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Johnson, MD, Study Chair — Mayo Clinic; Aaron Mansfield, MD, Principal Investigator — Mayo Clinic, Rochester, MN; Mitesh J Borad, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota